CLINICAL TRIAL: NCT01211392
Title: Detection of Bone Marrow Changes: Comparison of MRI and DECT
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Gustav Andreisek, MD, University of Zurich
Other Study IDs: 005
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Bone Marrow Changes
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Other: magnetic resonance imaging — magnetic resonance imaging is compared to dual-energy computed tomography for the detection of bone marrow changes

SUMMARY:
Prospective study where magnetic resonance imaging is compared to dual-energy computed tomography for the detection of bone marrow changes.

ELIGIBILITY:
Inclusion criteria:

* Patients with bone marrow changes

Exclusion criteria:

* Pregnacy
* Age below 18 ys old
* Contraindications for MRI

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bone marrow changes
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland